CLINICAL TRIAL: NCT06787079
Title: Effect of Kinesio Taping Application in Addition to Pilates Exercises on Core Muscle Thickness, Cognition and Mental Fatigue in Individuals With Non-specific Low Back Pain: A Randomized Placebo-Controlled Study
Brief Title: Effect of Kinesio Taping Application in Addition to Pilates Exercises on Core Muscle Thickness, Cognition and Mental Fatigue in Individuals With Non-specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ilayda Dilan Isik, Msc, Physiotherapist, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AnkaraSBU
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain; Non Specific Low Back Pain
Keywords: low back pain; kinesio tape; pilates; core; cognition; mental fatigue
MeSH Terms: conditions — Low Back Pain; Mental Fatigue | interventions — Athletic Tape; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Tape and Pilates Group (Active Comparator): Kinesio taping will be applied to this group in addition to the Pilates exercise protocol.
  Interventions: Other: Kinesio Tape; Other: Pilates
- Placebo Tape and Pilates Group (Placebo Comparator): Flaster taping will be applied to this group in addition to the Pilates exercise protocol.
  Interventions: Other: Pilates; Other: Placebo
- Pilates Group (Other): Only the Pilates exercise protocol will be applied to this group.
  Interventions: Other: Pilates

INTERVENTIONS:
Other: Kinesio Tape — Kinesio tape is a non-invasive therapeutic approach that does not involve any medication. It is often used to support tissue and reduce pain.
  Arms: Kinesio Tape and Pilates Group
Other: Pilates — Pilates exercises are mind-body exercises that are performed on a mat or with special equipment and focus on strength, core stability, flexibility, muscle control, posture and breathing. Pilates exercises are frequently used to develop elements such as core stability, muscle flexibility and strength, physical fitness and body awareness.
Other: Placebo — Placebo taping will be applied in the same way as kinesio taping, but with plaster tape.
  Arms: Placebo Tape and Pilates Group

SUMMARY:
Low back pain is a common problem. In low back pain, the core region and posture are frequently affected. However, no definitive decision has been reached regarding cognition and mental fatigue. In the treatment of low back pain, exercise and kinesio taping approaches are frequently used. The aim of this study is to evaluate the effects of kinesio taping applied in addition to pilates exercises on pain, core muscle thickness, strength and endurance, posture, cognition and mental fatigue in individuals with non-specific low back pain and to compare it with placebo taping and the control group. The primary outcome measure of this study is core muscle thickness, while other measurements will be considered as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Having back pain of at least 3 out of 10 points on the Visual Analog Scale,

  * Being between the ages of 30-55,
  * Having back pain for at least 1 month,
  * Having been tested with a test piece beforehand and not having an allergy to kinesio taping.

Exclusion Criteria:

* • Having had surgery for back pain,

  * Not complying with treatment,
  * Having a neurological deficit,
  * Having a body mass index over 30,
  * Having a positive straight leg raising test,
  * Having a positive slump test,
  * Having a positive bowstring test,
  * Being pregnant,
  * Having received any treatment for back pain in the last month,
  * Doing regular exercise in the last month.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Core Muscle Thickness | Beginning, Week 3, Week 6
  Core muscle thickness will be measured with ultrasound. The measurement will be taken first in the resting position and then by performing the hollowing maneuver. The difference between the two will be recorded.

SECONDARY OUTCOMES:
Pain | Beginning, Week 3, Week 6
  Visual analog scale (VAS) will be used in pain assessment. Patients will be asked to mark the pain intensity on a 10 cm scale defined as "0 (no pain)" and "10 (unbearable pain)". The point marked on the scale will be measured with a ruler (in cm) and recorded. Pain intensity will be evaluated in three different situations: activity, rest and night pain.
Core Muscle Strength | Beginning, Week 3, Week 6
  A pressurized biofeedback unit (BBU) will be used when evaluating muscle strength. BBU is a device that can be used to measure muscle function by detecting the movement of a muscle. Before the measurement, the person will be taught the "Abdominal Hollowing" maneuver, which is a maneuver to pull the abdominal wall inward by saying "Pull your belly up and in." Then, while the person is lying face down, the device will be fixed at 70mmHg and placed at the person's anterior superior iliac level. Then, the person will be asked to perform the maneuver and continue it for 10 seconds, and the change in pressure will be recorded. It will be repeated 3 times and the best measurement will be taken as the final measurement.
Core Muscle Endurance | Beginning, Week 3, Week 6
  The endurance of the core muscles will be evaluated in plank and side plank positions. Individuals will be asked to stand in plank and bilateral side plank positions and how long they can maintain this position will be measured.
Posture | Beginning, Week 3, Week 6
  The "APECS (AI Posture Evaluation and Correction System)" mobile application will be used in posture assessment. For measurements, photographs will be taken from the front and side and analyzed with the program. The degrees given by the analysis will be noted on the assessment form and comparison will be made.
Cognition | Beginning, Week 3, Week 6
  Montreal Cognitive Assessment will be used in cognition assessment. The maximum score for this scale is 30. 21 and above is considered good.
Mental Fatigue | Beginning, Week 3, Week 6
  The Mental Fatigue Scale (MFS) will be used when assessing mental fatigue. The MFS was created to measure the effects of mental fatigue in various life situations. The person will be asked to answer the scale questions and then the score for each question will be added up. The higher the total score, the higher the mental fatigue is reported to be. The maximum score can be 38.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Sağlık Bilimleri Üniversitesi, Ankara
  - GYM Center, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sheng Y, Duan Z, Qu Q, Chen W, Yu B. Kinesio taping in treatment of chronic non-specific low back pain: a systematic review and meta-analysis. J Rehabil Med. 2019 Oct 29;51(10):734-740. doi: 10.2340/16501977-2605. PMID 31544952
- [Background] Eliks M, Zgorzalewicz-Stachowiak M, Zenczak-Praga K. Application of Pilates-based exercises in the treatment of chronic non-specific low back pain: state of the art. Postgrad Med J. 2019 Jan;95(1119):41-45. doi: 10.1136/postgradmedj-2018-135920. Epub 2019 Jan 12. PMID 30636192
- [Background] Ogunniran IA, Akodu AK, Odebiyi DO. Effects of kinesiology taping and core stability exercise on clinical variables in patients with non-specific chronic low back pain: A randomized controlled trial. J Bodyw Mov Ther. 2023 Jan;33:20-27. doi: 10.1016/j.jbmt.2022.09.013. Epub 2022 Sep 28. PMID 36775519
- See also: MoCA usage permission and the Turkish version of the survey were taken from this page. — https://mocacognition.com/